CLINICAL TRIAL: NCT00981721
Title: A Phase I, Randomised, Multi-centre, Open-label Study to Determine the Pharmacokinetics and Tolerability of Cediranib (RECENTIN™, AZD2171) Following a Single and Multiple Oral 20mg or 30 mg Doses in Chinese Patients With Advanced Solid Malignancies
Brief Title: A Study to Determine the Pharmacokinetics of Cediranib in Chinese Patients With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8480C00060
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2011-06

CONDITIONS: Advanced Solid Malignancies
Keywords: Phase I; Advanced solid malignancies; Advanced solid tumour; Advanced cancer; Cediranib (RECENTIN™, AZD2171); China; PK; pharmacokinetics
MeSH Terms: interventions — cediranib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): cediranib 20mg
  Interventions: Drug: cediranib (RECENTIN TM, AZD2171)
- 2 (Experimental): cediranib 30mg
  Interventions: Drug: cediranib (RECENTIN TM, AZD2171)

INTERVENTIONS:
Drug: cediranib (RECENTIN TM, AZD2171) — 20 mg or 30mg cediranib once on Days 1, then 20 mg or 30mg cediranib once daily from Days 8

SUMMARY:
This study is being carried out to see how single and multiple doses of cediranib are handled by the body (that is how they are absorbed, broken down and got rid of from the body) by measuring levels of drug in the blood in Chinese patients with advanced solid malignancies.

The study will also assess the tolerability of 20 or 30 mg cediranib in Chinese patients and how the tumour responds to treatment with cediranib.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Histological and/or cytological confirmed advanced solid malignancies
* Refractory to conventional therapeutic modalities, or for which no appropriate therapies exist

Exclusion Criteria:

* For the first question: Patients with a history of poorly controlled hypertension with resting blood pressure >150/100 mmHg in the presence or absence of a stable regimen of antihypertensive therapy, or patients who are requiring maximal doses of calcium channel blockers to stabilize blood pressure.
* Significant haemorrhage (>30 ml/bleeding episode in previous 3 months), haemoptysis (>5 ml fresh blood in previous 4 weeks) or thrombotic event (including transient ischaemic attack) in the previous 12 months
* Recent(<28 days) major thoracic and abdominal surgery prior to entry into the study, or a surgical incision that is not fully healed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2010-05 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To assess the pharmacokinetics of single dose of cediranib 20mg or 30 mg by assessment of area under the curve over the time (AUC) and maximum concentration in Chinese patients with advanced solid malignant tumours | Multiple assessments in the first 6 days

SECONDARY OUTCOMES:
To assess the pharmacokinetics of multiple doses of cediranib 20mg or 30 mg in Chinese patients with advanced solid malignant tumours | Multiple assessments up to day 29
To assess the safety and tolerability of single and multiple doses of cediranib 20mg or 30 mg in Chinese patients with advanced solid malignancies. | Safety assessments to be taken until Day 29 (while patient remains on study treatment), then every 4 weeks until treatment discontinuation and then 30 day follow up

CONTACTS AND LOCATIONS:
Overall Officials: Jeannie Hou, Study Director — AstraZeneca China MC; Sun Yan, Prof, Principal Investigator — Cancer Hospital, CAMS&PUMC, China
Locations (2):
- China (2):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Hong Kong, Hong Kong